CLINICAL TRIAL: NCT04511429
Title: COVID-19 in Immunosuppressed Children
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: D'Or Institute for Research and Education (Other)
Collaborators: Hospital Estadual da Criança (Unknown); Hospital Federal de Bonsucesso (Other); Rio de Janeiro State Research Supporting Foundation (FAPERJ) (Other Government)
Responsible Party: Sponsor
Other Study IDs: 062-2020
Record Dates: First submitted 2020-07-24; First posted 2020-08-13 (Actual); Last update posted 2020-08-13 (Actual); Status verified 2020-08

CONDITIONS: Infections, Coronavirus; Kidney Transplantation; Liver Transplantation; Cancer; Covid19
Keywords: COVID-19; Kidney transplantation; Liver transplantation; Cancer; Children; Adolescents; Pediatrics
MeSH Terms: conditions — Coronavirus Infections; Neoplasms; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Kidney transplant patients: Patients submitted to kidney transplantation.
- Liver transplant patients: Patients submitted to liver transplantation.
- Oncological patients: Oncological patients submitted to chemotherapy.

SUMMARY:
Viral respiratory infections are common infectious complications after kidney transplantation, especially in the pediatric age group, and immunosuppressed patients may develop more severe disease. Immunosuppressive medications alter the patient's immune response by acting on humoral, cellular immunity and neutrophil function, increasing the risk of serious viral infections. Little is known about how these patients respond to infection by the new coronavirus (SARS-CoV-2).

Experience with SARS caused by the Influenza H1N1 virus suggests that the severity of the disease depends on pre-existing comorbidities and the individual immune response. In more severe cases, an imbalance between the inflammatory system and the immune system is observed, determining direct consequences when pro and anti-inflammatory cytokines reach the systemic circulation in an exacerbated and unbalanced manner. Such fact can generate "cytokine storm syndrome", resulting in multiple organ dysfunction syndrome.

March 2020 reports from Papa Giovanni XXIII Hospital in Bergamo, Italy - one of the largest pediatric liver transplant centers - showed that the number of transplant patients infected with Coronavirus disease 2019 (COVID- 19) increased progressively. However, they did not see greater severity and complications in this population. Immunosuppression could act as a protective factor.

The present study aims to describe the prevalence of viral infection by SARS-CoV-2 in a sample of immunosuppressed children, from three groups: kidney transplants, liver transplants and oncohematological. The investigators will also look for the epidemiological profile and clinical evolution of these patients, enabling a better understanding of the COVID-19 in this special population. The investigators' hypothesis is that infection with the new coronavirus may be asymptomatic in a large number of children and that immunosuppression, observed in liver and kidney transplant patients and also seen in cancer patients, may act as protection for severe forms of COVID-19.

After obtaining written informed consent from the family, the investigators will include patients from 0-18 years of age, on regular outpatient follow-up, symptomatic or not, and will check for the presence of IgM/IgG antibodies against the SARS-CoV-2. For those symptomatic or with a positive IgM result, material (oro/nasopharyngeal swabs) for RT-PCR trial for the new coronavirus will be collected. Demographic and clinical variables will be registered. The outcomes are: Serology for COVID-19 result; PCR for COVID-19 result; presence of symptoms of COVID-19; proportion of patients with viral shedding on days 3,7,14,21 and 30 after diagnosis; need for hospital admission; need for Intensive care admission; death.

DETAILED DESCRIPTION:
Variables to be measured

* Demographic data (initials, record, age, sex, race / ethnicity, weight, height, BMI).
* Epidemiological data:

  * For kidney transplant patients: time of transplant, in years and complete months; primary kidney disease; presence and time of onset of respiratory symptoms, in days; presence of risk factors or comorbidities; current immunosuppression (drugs and doses); serum level of calcineurin inhibitor on the day of collection; previous vaccination for Influenza; previous viral infections; date of the last episode of rejection treated.
  * For liver transplant patients: time of transplant, in years and complete months; primary liver disease; presence and time of onset of respiratory symptoms, in days; presence of risk factors or comorbidities; current immunosuppression (drugs and doses); serum level of calcineurin inhibitor on the day of collection; previous vaccination for Influenza; previous viral infections; date of the last episode of rejection treated.
  * For oncohematological patients: time of diagnosis, in years and complete months; primary oncohematological disease; treatment received for the oncohematological disease; presence and time of onset of respiratory symptoms, in days; presence of risk factors or comorbidities; current cancer treatment; previous vaccination for Influenza; previous viral infections.
* Clinics visit / hospitalization data: clinical picture: syndromic diagnosis / signs and symptoms; initial image exam: chest X-ray and / or chest CT; Treatment performed: antiviral, antibiotic, corticoid (reason / dose / time); respiratory support (oxygen therapy only / Non-Invasive Ventilation / High Flow Nasal Cannula / invasive mechanical pulmonary ventilation / ECMO - time of use (days); days free of oxygen therapy, Non-Invasive Ventilation and invasive mechanical pulmonary ventilation.
* Diagnosis of SARS-CoV-2 infection: rapid test for Covid-19 in the blood: IgM / IgG; rapid test for COVID-19 in nasopharyngeal or tracheal secretion.
* Outcomes: Serology for COVID-19 result; PCR for COVID-19 result; presence of symptoms of COVID-19; proportion of patients with viral shedding on days 3,7,14,21 and 30 after diagnosis; need for hospital admission; need for Intensive care admission; death.

ELIGIBILITY:
Inclusion Criteria:

* Renal or liver transplant patients, with functioning graft and using immunosuppression, in outpatient follow-up or hospitalized.
* Patients treating oncohematological disorders, in outpatient follow-up or hospitalized..

Exclusion Criteria:

* Patients who or whose parents refuse to sign the Informed Consent Form.

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients aged 0-18 years, immunosuppressed, kidney or liver transplanted, or oncologic patients, in outpatient follow-up or hospitalized.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-06-30 (Actual); Primary Completion 2020-10 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Serology (IgM, IgG) for COVID-19. | 9 months
  percentage of positivity

SECONDARY OUTCOMES:
Hospital admission | 9 months
  percentage of patients admitted to hospital
Intensive care admission | 9 months
  percentage of patients admitted to intensive care unit
Death | 9 months
  percentage of patients who died
Positive PCR for COVID-19 | 9 months
  percentage of positivity
Clinical characteristics of patients with COVID-19 | 9 months
  Percentage of patients with symptoms of COVID-19
Proportion of patients with viral excretion in respiratory secretion and faeces on days 3, 7, 14, 21 and 30 after confirmation of covid 19. | 9 months
  Percentage of patients with positive PCR in respiratory secretion and feces on days 3, 7, 14, 21 and 30 after confirmation of covid 19.

CONTACTS AND LOCATIONS:
Overall Officials: Thais L Cleto-Yamane, MD, MSc, Principal Investigator — D'Or Institute for Research and Education (IDOR); Arnaldo Prata-Barbosa, MD, PhD, Study Director — D'Or Institute for Research and Education (IDOR); Antonio José L A da Cunha, MD, PhD, Study Chair — Universidade Federal do Rio de Janeiro
Locations (2):
- Brazil (2):
  - Hospital Federal de Bonsucesso, Rio de Janeiro, Rio de Janeiro
  - Hospital Estadual da Criança, Rio de Janeiro, Rio de Janeiro

REFERENCES:
- [Result] Danziger-Isakov L, Steinbach WJ, Paulsen G, Munoz FM, Sweet LR, Green M, Michaels MG, Englund JA, Murray A, Halasa N, Dulek DE, Madan RP, Herold BC, Fisher BT. A Multicenter Consortium to Define the Epidemiology and Outcomes of Pediatric Solid Organ Transplant Recipients With Inpatient Respiratory Virus Infection. J Pediatric Infect Dis Soc. 2019 Jul 1;8(3):197-204. doi: 10.1093/jpids/piy024. PMID 29538674
- [Result] Lee KH, Yoo SG, Cho Y, Kwon DE, La Y, Han SH, Kim MS, Choi JS, Kim SI, Kim YS, Min YH, Cheong JW, Kim JS, Song YG. Characteristics of community-acquired respiratory viruses infections except seasonal influenza in transplant recipients and non-transplant critically ill patients. J Microbiol Immunol Infect. 2021 Apr;54(2):253-260. doi: 10.1016/j.jmii.2019.05.007. Epub 2019 Jun 19. PMID 31262511
- [Result] D'Antiga L. Coronaviruses and Immunosuppressed Patients: The Facts During the Third Epidemic. Liver Transpl. 2020 Jun;26(6):832-834. doi: 10.1002/lt.25756. Epub 2020 Apr 24. No abstract available. PMID 32196933
- [Result] Cortiula F, Pettke A, Bartoletti M, Puglisi F, Helleday T. Managing COVID-19 in the oncology clinic and avoiding the distraction effect. Ann Oncol. 2020 May;31(5):553-555. doi: 10.1016/j.annonc.2020.03.286. Epub 2020 Mar 19. No abstract available. PMID 32201224
- [Result] Ronco C, Reis T, De Rosa S. Coronavirus Epidemic and Extracorporeal Therapies in Intensive Care: si vis pacem para bellum. Blood Purif. 2020;49(3):255-258. doi: 10.1159/000507039. Epub 2020 Mar 13. No abstract available. PMID 32172242
- [Result] Memoli MJ, Athota R, Reed S, Czajkowski L, Bristol T, Proudfoot K, Hagey R, Voell J, Fiorentino C, Ademposi A, Shoham S, Taubenberger JK. The natural history of influenza infection in the severely immunocompromised vs nonimmunocompromised hosts. Clin Infect Dis. 2014 Jan;58(2):214-24. doi: 10.1093/cid/cit725. Epub 2013 Nov 1. PMID 24186906
- [Result] Fitzner J, Qasmieh S, Mounts AW, Alexander B, Besselaar T, Briand S, Brown C, Clark S, Dueger E, Gross D, Hauge S, Hirve S, Jorgensen P, Katz MA, Mafi A, Malik M, McCarron M, Meerhoff T, Mori Y, Mott J, Olivera MTDC, Ortiz JR, Palekar R, Rebelo-de-Andrade H, Soetens L, Yahaya AA, Zhang W, Vandemaele K. Revision of clinical case definitions: influenza-like illness and severe acute respiratory infection. Bull World Health Organ. 2018 Feb 1;96(2):122-128. doi: 10.2471/BLT.17.194514. Epub 2017 Nov 27. PMID 29403115
- [Result] Kumar D, Tellier R, Draker R, Levy G, Humar A. Severe Acute Respiratory Syndrome (SARS) in a liver transplant recipient and guidelines for donor SARS screening. Am J Transplant. 2003 Aug;3(8):977-81. doi: 10.1034/j.1600-6143.2003.00197.x. PMID 12859532
- [Result] Liang W, Guan W, Chen R, Wang W, Li J, Xu K, Li C, Ai Q, Lu W, Liang H, Li S, He J. Cancer patients in SARS-CoV-2 infection: a nationwide analysis in China. Lancet Oncol. 2020 Mar;21(3):335-337. doi: 10.1016/S1470-2045(20)30096-6. Epub 2020 Feb 14. No abstract available. PMID 32066541

DOCUMENTS (2):
  • Informed Consent Form (2020-07-01): https://cdn.clinicaltrials.gov/large-docs/29/NCT04511429/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2020-07-01): https://cdn.clinicaltrials.gov/large-docs/29/NCT04511429/Prot_SAP_001.pdf